CLINICAL TRIAL: NCT02629666
Title: Exercise Referral Schemes Enhanced by Self-Management Strategies to Battle Sedentary Behaviour
Acronym: SitLESS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ramon Llull (Other)
Collaborators: Fundació Salut i Envelliment de la Universitat Autònoma de Barcelona (Unknown); University of Southern Denmark (Other); Queen's University, Belfast (Other); University of Ulm (Other); Sport Initiative et Loisir Bleu Association (Unknown); University of Glasgow (Other)
Responsible Party: Principal Investigator, Dra. Maria Giné Garriga, Professor (PT, PhD), University Ramon Llull
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PHC-17-2014. 634270-2.
Record Dates: First submitted 2015-11-19; First posted 2015-12-14 (Estimated); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Physical Activity; Biological Aging; Frail Older Adults; Controlled Clinical Trials, Randomized; Sedentary Behaviour; Exercise Referral Schemes; Physical Function
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Exercise Referral Scheme (ERS) (Active Comparator): In the Exercise Referral Scheme (ERS) intervention participants will undergo a physical activity program of 16 weeks, with two sessions per week (60 minutes each session). Participants will be asked to perform the activity in a moderate to vigorous intensity (according to each individual's progression) during the central part of each session. Intensity will be estimated using the modified Borg Scale of Perceived Exertion (e.g. moderate intensity activity will be considered as a 4 to 6 and vigorous-intensity activity as a 7 to 9) or with training loads (i.e. ankle weights and dumbbells) corresponding to 70-80% of maximum, adjusted progressively during the training period. ERS programs will be based on a combination of aerobic, strength-based, balance and flexibility activities, with a specially trained PA specialist. These sessions will be always performed under the supervision of the same trainer. The PA intervention is adapted to the participants' functional status.
  Interventions: Behavioral: ERS and/or Self-management Strategies
- ERS + Self-management Strategies (Experimental): Participants will undergo the aforementioned Physical Activity program plus 11 sessions of Self-Management Strategies (SMS).
  SMS start with a face-to-face session in an indoor primary-care facility. The next 6 sessions are further implemented in a group format. SMS are aimed at increasing self-efficacy in reducing sedentary behaviour and at adopting/maintaining an active behaviour as complement to a standard physical activity program (ERS). SMS group sessions will be conducted during week 3 to 11 of the ERS, after the PA sessions (6 sessions: 3 once a week, 3 once every second week). There will be 4 telephone contacts during the adherence phase, at week 15, 20, 25 and 30.
  Interventions: Behavioral: ERS and/or Self-management Strategies
- Control group (No Intervention): Researchers will give to all participants during the first informative meeting (prior assessment) a written general booklet standardized across sites with WHO recommendation regarding PA regular practice for health. During the intervention, a health advice meeting with standardized topics about healthy lifestyle and feedback on some outcomes regarding their results will be held twice in the Primary Health Centre (at week 5, and at week 11). Researchers will send a letter or phone call prior to each follow up reminding the next assessment.

INTERVENTIONS:
Behavioral: ERS and/or Self-management Strategies
  Arms: ERS + Self-management Strategies; Exercise Referral Scheme (ERS)

SUMMARY:
The increase of the elderly population leads to increased prevalence of frailty, risk for poor health outcomes, and related health and social care costs. Lack of physical activity (PA) and established sedentary behaviours (SB) constitute an additional burden, as they are related to progression of chronic disease and disabling conditions. An existing initiative to battle SB and insufficient PA levels are exercise referral schemes (ERS) implemented in primary care, where insufficiently active individuals are referred to a third party service (sports centre or leisure facility) that prescribes and monitors an exercise programme tailored to the patients' needs. ERS had shown improvements in PA in the short-term, but may have limited power to change SB and produce long-term effects. Thus, ERS might be enhanced by self-management strategies (SMS) to promote behavioural change. Such strategies based on social cognitive theory have been shown to increase self-confidence, power to act, and involvement in exercise. In a first stage, a systematic review, focus groups and a feasibility study will be conducted. Then, a three-armed pragmatic randomized controlled trial (RCT) will assess the long-term effectiveness (18-month follow-up) of a complex intervention on sedentary behaviour (SB) in an elderly population, based on existing ERS enhanced by self-management strategies (SMS). It will be compared to ERS alone and to general recommendations plus two educational sessions. The RCT will include 1338 subjects and will have a follow up of 18 months. The effect on SB will be measured as sitting time and the number of minutes spent in activities requiring ≤ 1.5 Metabolic Equivalent Tasks, and PA as daily counts per minute and intensity of exercise, and daily step counts. Secondary outcomes will include: physical function, healthcare use and costs, anthropometry, bioimpedance, blood pressure, self-rated health and quality of life, activities of daily living, anxiety, depressive symptoms, social network, physical activity self-regulation, self-efficacy for exercise, disability, fear of falling, loneliness, executive function, and physical fatigue. In a subsample, the level of frailty-associated biomarkers and inflammation, and sarcopenia-associated markers of muscle quality will be analysed. A process evaluation will be performed throughout the trial. SITLESS will assess policy makers in deciding how or whether ERS should be further implemented or restructured in order to increase its adherence, efficacy and cost-effectiveness.

ELIGIBILITY:
Inclusion Criteria:

Community-dwelling older persons aged 65 or above.

Able to walk without help of another person during 2 minutes, and without major physical limitations, defined as a score on the Short Physical Performance Battery (Guralnik et al., 1995) of 4 or above. The use of an assistive device will be permitted.

Insufficiently active and/or Self-report sitting too much during a usual day. Answer yes to the following question: 'Do you perform regular physical activity (PA) at least 30 minutes five or more days of the week (please only refer to physical activity that makes the participant run out of breath while doing it or it doesn't allow him/her to maintain a conversation while doing the activity (do not count regular walking)?'

And/or answer yes to question: 'For most days, do you feel you sit for too long (6-8 hours or more a day)? Some examples might include when watching TV, working the computer / laptop or when doing sitting-based hobbies such as sewing'.

Exclusion Criteria:

Dementia assessed with the six-Item Screener. Participants with three or more errors should be excluded.

Unstable medical conditions (e.g. elevated blood pressure after medication) or with symptomatic cardiovascular disease.

Any medical condition which may interfere with the study design (e.g. end-stage disease).

Refuse to wear an accelerometer (primary outcome)

Unable to attend during the study period (80% of the total sessions).

Had participated in an ERS in the 6 months prior the study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 1360 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2020-02 (Actual)

PRIMARY OUTCOMES:
Change in sitting time | During 7 days. Outcome measure will be collected (T0) baseline pre-intervention, (T1) at month 4 post intervention, (T2) at month 16 (12 months after the end of the intervention), and (T3) at month 22 (18 months after the end of the intervention)
  Sitting time with activity monitors (Actigraph, Axivity, ActivPal) (minutes) and with Sedentary Behavior Questionnaire.
Change in minutes spent in sedentary behaviour | During 7 days. Outcome measure will be collected (T0) baseline pre-intervention, (T1) at month 4 post intervention, (T2) at month 16 (12 months after the end of the intervention), and (T3) at month 22 (18 months after the end of the intervention)
  Number of minutes spent in activities requiring ≤ 1.5 Metabolic Equivalent Tasks with Actigraph activity monitor.
Change in total activity counts per minute | During 7 days. Outcome measure will be collected (T0) baseline pre-intervention, (T1) at month 4 post intervention, (T2) at month 16 (12 months after the end of the intervention), and (T3) at month 22 (18 months after the end of the intervention)
  Daily counts per minute with Actigraph activity monitor.

SECONDARY OUTCOMES:
Change in use and costs of the healthcare system | Outcome measure will be collected (T0) baseline pre-intervention, (T1) at month 4 post intervention, (T2) at month 16 (12 months after the end of the intervention), and (T3) at month 22 (18 months after the end of the intervention)
  Use of sport services, and use of health and social services, medications, number of falls.
Change in % fat and % muscle | Outcome measure will be collected (T0) baseline pre-intervention, (T1) at month 4 post intervention, (T2) at month 16 (12 months after the end of the intervention), and (T3) at month 22 (18 months after the end of the intervention)
  Tanita BC 420S MA bioimpedance analyser.
Change in health-related quality of life | Outcome measure will be collected (T0) baseline pre-intervention, (T1) at month 4 post intervention, (T2) at month 16 (12 months after the end of the intervention), and (T3) at month 22 (18 months after the end of the intervention)
  SF-12 (units), EUROQOL-5D, and ICECAP-O questionnaires.
Change in activities of daily living performance | Outcome measure will be collected (T0) baseline pre-intervention, (T1) at month 4 post intervention, (T2) at month 16 (12 months after the end of the intervention), and (T3) at month 22 (18 months after the end of the intervention)
  6-item questionnaire (Saliba et al., 2000).
Change in depressive symptoms | Outcome measure will be collected (T0) baseline pre-intervention, (T1) at month 4 post intervention, (T2) at month 16 (12 months after the end of the intervention), and (T3) at month 22 (18 months after the end of the intervention)
  Hospital Anxiety and Depression Scale
Change in anxiety symptoms | Outcome measure will be collected (T0) baseline pre-intervention, (T1) at month 4 post intervention, (T2) at month 16 (12 months after the end of the intervention), and (T3) at month 22 (18 months after the end of the intervention)
  Hospital Anxiety and Depression Scale
Changes in social network | Outcome measure will be collected (T0) baseline pre-intervention, (T1) at month 4 post intervention, (T2) at month 16 (12 months after the end of the intervention), and (T3) at month 22 (18 months after the end of the intervention)
  Lubben Social Network Scale-6
Changes in Physical activity self-regulation | Outcome measure will be collected (T0) baseline pre-intervention, (T1) at month 4 post intervention, (T2) at month 16 (12 months after the end of the intervention), and (T3) at month 22 (18 months after the end of the intervention)
  12-item Physical Activity Self-Regulation Scale
Changes in Self-efficacy for exercise | Outcome measure will be collected (T0) baseline pre-intervention, (T1) at month 4 post intervention, (T2) at month 16 (12 months after the end of the intervention), and (T3) at month 22 (18 months after the end of the intervention)
  Marcus's Self-Efficacy Questionnaire
Changes in Disability | Outcome measure will be collected (T0) baseline pre-intervention, (T1) at month 4 post intervention, (T2) at month 16 (12 months after the end of the intervention), and (T3) at month 22 (18 months after the end of the intervention)
  Short form Late Life Function and Disability Index
Changes in Fear of falling | Outcome measure will be collected (T0) baseline pre-intervention, (T1) at month 4 post intervention, (T2) at month 16 (12 months after the end of the intervention), and (T3) at month 22 (18 months after the end of the intervention)
  Short Falls Efficacy Scale - International
Change in Loneliness perception | Outcome measure will be collected (T0) baseline pre-intervention, (T1) at month 4 post intervention, (T2) at month 16 (12 months after the end of the intervention), and (T3) at month 22 (18 months after the end of the intervention)
  Short form De Jong Gierveld Loneliness Scale
Change in Executive function | Outcome measure will be collected (T0) baseline pre-intervention, (T1) at month 4 post intervention, (T2) at month 16 (12 months after the end of the intervention), and (T3) at month 22 (18 months after the end of the intervention)
  Trail Making Test
Change in Physical fatigue | Outcome measure will be collected (T0) baseline pre-intervention, (T1) at month 4 post intervention, (T2) at month 16 (12 months after the end of the intervention), and (T3) at month 22 (18 months after the end of the intervention)
  Pittsburg Fatigability Scale
Change in general function | Outcome measure will be collected (T0) baseline pre-intervention, (T1) at month 4 post intervention, (T2) at month 16 (12 months after the end of the intervention), and (T3) at month 22 (18 months after the end of the intervention)
  Short Physical Performance Battery
Change in handgrip strength | Outcome measure will be collected (T0) baseline pre-intervention, (T1) at month 4 post intervention, (T2) at month 16 (12 months after the end of the intervention), and (T3) at month 22 (18 months after the end of the intervention)
  Takei analogue Hand Grip Dynamometer
Change in aerobic capacity | Outcome measure will be collected (T0) baseline pre-intervention, (T1) at month 4 post intervention, (T2) at month 16 (12 months after the end of the intervention), and (T3) at month 22 (18 months after the end of the intervention)
  2-minutes' walk test
Change in static balance | Outcome measure will be collected (T0) baseline pre-intervention, (T1) at month 4 post intervention, (T2) at month 16 (12 months after the end of the intervention), and (T3) at month 22 (18 months after the end of the intervention)
  Unipedal stance
Change in mean strength and power with concentric contraction of isoinertial movement | Outcome measure will be collected (T0) baseline pre-intervention, (T1) at month 4 post intervention, (T2) at month 16 (12 months after the end of the intervention), and (T3) at month 22 (18 months after the end of the intervention)
  Linear encoder in 3 activities of daily living with: (a) 30-second chair stand rise; (b) five repetitions of arm curl with both hands with a 2-kg weight; and (c) four counter-movement jumps.

OTHER OUTCOMES:
Level of frailty-associated biomarkers and inflammation | Outcome measure will be collected (T0) baseline pre-intervention, and (T1) at month 4 post intervention
  Blood sample: IL-6, hsCRP, TNF-alpha, IGF-1.
Sarcopenia-associated markers of muscle quality | Outcome measure will be collected (T1) at month 4 post intervention
  Muscle biopsy: Myostatin, IL-6, IL-8, IL-15, VEGF, BDNF, FGF21, irisin, Type 2/Type 1 fibre ratio, Wnt and Notch signaling, CDC42.

CONTACTS AND LOCATIONS:
Locations (1):
- Facultat de Psicologia, Ciències de l'Educació i de l'Esport Blanquerna, Barcelona, Please Select, Spain

REFERENCES:
- [Derived] Svensson NH, Thorlund JB, Ollgaard Olsen P, Sondergaard J, Wehberg S, Andersen HS, Caserotti P, Thilsing T. Effect of exercise referral schemes and self-management strategies on healthcare service utilisation among community-dwelling older adults: secondary analyses of two randomised controlled trials. BMJ Open. 2024 Nov 2;14(11):e084938. doi: 10.1136/bmjopen-2024-084938. PMID 39488430
- [Derived] Drahota A, Udell JE, Mackenzie H, Pugh MT. Psychological and educational interventions for preventing falls in older people living in the community. Cochrane Database Syst Rev. 2024 Oct 3;10(10):CD013480. doi: 10.1002/14651858.CD013480.pub2. PMID 39360568
- [Derived] Bizjak DA, Zugel M, Schumann U, Tully MA, Dallmeier D, Denkinger M, Steinacker JM. Do skeletal muscle composition and gene expression as well as acute exercise-induced serum adaptations in older adults depend on fitness status? BMC Geriatr. 2021 Dec 15;21(1):697. doi: 10.1186/s12877-021-02666-0. PMID 34911479
- [Derived] Coll-Planas L, Blancafort Alias S, Tully M, Caserotti P, Gine-Garriga M, Blackburn N, Skjodt M, Wirth K, Deidda M, McIntosh E, Rothenbacher D, Gallardo Rodriguez R, Jerez-Roig J, Sansano-Nadal O, Santiago M, Wilson J, Guerra-Balic M, Martin-Borras C, Gonzalez D, Lefebvre G, Denkinger M, Kee F, Salva Casanovas A, Roque I Figuls M; SITLESS group. Exercise referral schemes enhanced by self-management strategies to reduce sedentary behaviour and increase physical activity among community-dwelling older adults from four European countries: protocol for the process evaluation of the SITLESS randomised controlled trial. BMJ Open. 2019 Jun 14;9(6):e027073. doi: 10.1136/bmjopen-2018-027073. PMID 31203243
- [Derived] Deidda M, Coll-Planas L, Gine-Garriga M, Guerra-Balic M, Roque I Figuls M, Tully MA, Caserotti P, Rothenbacher D, Salva Casanovas A, Kee F, Blackburn NE, Wilson JJ, Skjodt M, Denkinger M, Wirth K, McIntosh E; SITLESS Team. Cost-effectiveness of exercise referral schemes enhanced by self-management strategies to battle sedentary behaviour in older adults: protocol for an economic evaluation alongside the SITLESS three-armed pragmatic randomised controlled trial. BMJ Open. 2018 Oct 15;8(10):e022266. doi: 10.1136/bmjopen-2018-022266. PMID 30327403
- [Derived] Gine-Garriga M, Coll-Planas L, Guerra M, Domingo A, Roque M, Caserotti P, Denkinger M, Rothenbacher D, Tully MA, Kee F, McIntosh E, Martin-Borras C, Oviedo GR, Jerez-Roig J, Santiago M, Sansano O, Varela G, Skjodt M, Wirth K, Dallmeier D, Klenk J, Wilson JJ, Blackburn NE, Deidda M, Lefebvre G, Gonzalez D, Salva A. The SITLESS project: exercise referral schemes enhanced by self-management strategies to battle sedentary behaviour in older adults: study protocol for a randomised controlled trial. Trials. 2017 May 18;18(1):221. doi: 10.1186/s13063-017-1956-x. PMID 28521831
- See also: SitLESS web page — http://www.sitless.eu